CLINICAL TRIAL: NCT07239154
Title: Clinical and Radiographic Assessment of Injectable Composite Versus Packable Composite in the Restoration of Cavitated Primary Molars a Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Injectable Composite Versus Packable Composite in Restoring of Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eslam samy abdel monaem kalboush (Other)
Responsible Party: Sponsor-Investigator, Eslam samy abdel monaem kalboush, Assistant lecturer in pediatric dentistry department delta university, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191131345021234567891911313450
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries in Children
Keywords: Decayed
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: outcome assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injectable composite (Experimental): it is a type of zero flow injectable composite used to restore teeth and molars
  Interventions: Other: injectable composite
- Packable composite (Other): composite used to restore molars
  Interventions: Other: packable composite

INTERVENTIONS:
Other: packable composite — packable composite used to restore teeth and molars
  Arms: Packable composite
Other: injectable composite — type of zero flow injectable composite
  Arms: injectable composite

SUMMARY:
This randomized clinical trial aims to compare the clinical and radiographic performance of injectable composite versus packable composite in restoring cavitated primary molars in children aged 4 to 8 years.

Study Purpose

To determine whether injectable composite performs as well as packable composite in Class I and II restorations in primary molars clinically and radiographically.

DETAILED DESCRIPTION:
This randomized clinical trial aims to compare the clinical and radiographic performance of injectable composite versus packable composite in restoring cavitated primary molars in children aged 4-8 years.

Study Purpose

To determine whether injectable composite performs as well packable composite in Class I and II restorations in primary molars.

Study Design

Type: Randomized clinical trial

Sample: 64 primary molars (32 per group)

Allocation: 1:1 using concealed envelopes

Group I (Experimental group): Injectable composite (Beautifil Flow Plus X F00, Shofu, Japan) Group II (Control group): Packable composite (Beautifil II LS, Shofu, Japan)

Follow-up: Clinical at 3, 6, 12 months

Radiographic at 0, 6, 12 months

Location: Pediatric Dentistry Clinic, Cairo University

Outcome Measures

Primary Outcome Clinical Performance (FDI Criteria):

Functional: marginal adaptation, fracture, proximal contact, occlusion, wear

Biological: caries at margins, hard tissue defects, sensitivity, pulp status

Esthetic: texture, staining, color match

Secondary Outcome Radiographic Performance:

Presence/absence of voids

Marginal integrity on bitewing radiographs

Rationale

Injectable composites may offer:

Better cavity adaptation

Easier handling

Shorter chair time (important in pediatric dentistry)

Packable composites offer:

Higher strength and wear resistance

The study investigates whether injectables can match or outperform packables clinically.

Hypothesis

Null hypothesis: There is no difference between injectable and packable composites in clinical and radiographic success.

Intervention The principal investigator ES will carry out all treatment procedures, and the patients will be randomly assigned to any of them.

For both groups:

1. Informed consent from participating children parents.
2. Baseline records photographs, percussion test, periapical radiograph and personal data collection (Appendix 1: Diagnostic chart).
3. Diagnostic chart with personal, medical and dental history will be filled (Appendix 1:

   Diagnostic chart).
4. Allocation (concealed by withdrawing a sealed opaque envelope containing Four-folded numbered papers containing the type of restorative material that will be used then writing the patient name and I.D. on it and will be opened after performing the cavity).
5. Clinical examination will be performed to assess the clinical inclusion criteria.
6. Preoperative and Postoperative photographs will be taken. 10
7. The radiographic examination will be performed by taking a periapical x-ray using (bitewing technique) to assess the inclusion criteria. The preoperative radiograph will serve as a reference for the follow-up radiographs.
8. Administration of local anesthesia at the side of the affected tooth.
9. Application of rubber dam for isolation, then caries removal procedure will be performed using a sterile round end bur in a high-speed hand piece and walls will be finished by a sterile fissure bur.
10. After cavity preparation, conditioning of the tooth will be done using phosphoric acid 35% for 30 seconds to enamel and 10 seconds for dentin then after rinsing the acid etch by water for 10 seconds bond will be applied to the tooth using bond brush then cured for 20 seconds.
11. The restorative material will be placed in the cavity and will be cured for 40 seconds.
12. The last step is to finish and polish the restoration material.
13. Clinical assessment will be done after each visit using FDI criteria to assess the clinical performance of each restoration in the three domains (biological, functional and aesthetics) and radiographic assessment will be done for 0, 6, and 12 months using preapical bitewing x-ray.

Sample size calculation:

Data will be analyzed using Medcalc software, version 22 for windows (MedCalc Software Ltd, Ostend, Belgium).

Categorical data will be described as frequency and percentage. Intergroup comparisons between categorical variables will be performed using the chi square test, while intragroup comparisons within each intervention will be performed using Cochran's Q test followed by pairwise multiple comparisons.

A p-value less than or equal to 0.05 will be considered statistically significant, and all tests will be two tailed. Statistical power of the study will be set at 80% with a 95% confidence level.

The sample size was calculated based on a previous study by Inthihas et al in 2019, in which the success rate of proximal giomer restorations in primary molars was 94.1% after 12 months (17).

By implementing a two tailed Z test for the difference between two independent proportions with an alpha level of 5% and a power of 80%.

The minimum sample size needed was 28 per group in order to detect a difference of 30%.

Sample size was increased by 15% to compensate for possible dropouts to reach 32 teeth per group. Sample size was performed using G*Power version 3.1.9.2 for windows.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Children aged 4-8 years.
  * Medically free.

Teeth:

* Restorable Class I and II cavities.
* Asymptomatic tooth.

Pre-operative radiographic examination:

* Absence of periapical or inter-radicular radiolucency.
* Absence of widening of periodontal ligaments space.
* Absence of internal or external root resorption.

Exclusion Criteria:

* Patients:

  * Uncooperative children.
  * Unable to attend follow-up visits.
  * Parents refuse to sign the informed consent.
  * Children participating in any other clinical trial involving fluoride therapy or other interventions that could directly influence caries development during the study period.

Teeth:

* Teeth which were previously restored.
* Mobility.

Pre-operative radiographic examination:

* Caries extending deep sub-gingivally.
* The tooth is about to exfoliate.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Assessment of Injectable Composite Versus Packable Composite in The Restoration of Cavitated Primary Molars | Time: T0 = baseline assessment and procedure will be done. T1 =3 months follow up. T2 = 6 months follow up. T3 = One-year follow-up.
  Clinical evaluation will be done according to Fédération Dentaire Internationale FDI criteria
  Scores:
  Clinically excellent = 1 Clinically good = 2 Clinically sufficient = 3 Clinically unsatisfactory = 4 Clinically poor = 5

SECONDARY OUTCOMES:
Radiographic Assessment of Injectable Composite Versus Packable Composite in The Restoration of Cavitated Primary Molars. | t = 0 months t2 = 6 months t3 = 12 months
  radiographic assessment will be done by using bitewing x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Eslam Kalboush, Mcs, Principal Investigator — Cairo University
Locations (1):
- faculty of dentistry,Cairo university, Cairo, Egypt